CLINICAL TRIAL: NCT03381807
Title: Human Amniotic Epithelial Stem Cell in Treatment of Refractory Severe Intrauterine Adhesion
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-080
Record Dates: First submitted 2017-11-27; First posted 2017-12-22 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCRA and intrauterine infusion of hAESCs (Experimental): hAESCs is infused into uterine cavity after TCRA.
  Interventions: Biological: hAESCs

INTERVENTIONS:
Biological: hAESCs — 5*10^7 hAESCs is infused into uterine cavity with TCRA on Day0, Day7 and after the first menstruation

SUMMARY:
This project will investigate the safety and effectiveness of human amniotic epithelial stem cells for treatment of severe refractory Asherman's syndrome.

DETAILED DESCRIPTION:
Asherman's syndrome is an gynecological disorder caused by the destruction of the endometrium due to repeated or aggressive curettages and/or endometritis. As a result, there is a loss of functional endometrium in multiple areas and the uterine cavity is obliterated by intrauterine adhesions, which results in amenorrhea, hypomenorrhea, infertility and recurrent pregnancy loss. Transcervical resection of adhesion (TCRA) is the main treatment for Asherman's syndrome; so far the effect is usually poor in moderate to severe refractory cases.

Human amniotic epithelial stem cells (hAESCs) are derived from human amniotic epithelium. hAESCs retain the characteristics approximating to embryonic stem cells. Animal experiments have shown that the endometrial thickness and fertility of mice was significantly improved after intrauterine therapy with hAESCs. To further explore the role of hAESCs in Asherman's syndrome patients, this project will evaluate the safety of hAESCs and find an effective treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

* 1. Previously diagnosed as uterine adhesion, after the operation of TCRA and the postoperatively standardized hormonal replacement therapy(HRT) , recently diagnosed with refractory Asherman's syndrome or endometrial atrophy(EA);
* 2. According to the American Fertility Society(AFS) classification in 1988, patients are diagnosed of AS or EA stageⅢ-Ⅳ confirmed by hysteroscopy;
* 3. Elimination of infertility, recurrent spontaneous abortion or hypomenorrhea caused by other diseases;
* 4. Be willing to maintain an HRT cycle medication throughout the study, unless it is not tolerated;
* 5. Normal blood coagulation, liver, heart, and kidney function, absence of HIV, Hepatitis B or C, syphilis and psychiatric pathology;
* 6. Be willing to complete the study and sign the consent form.

Exclusion Criteria:

* 1. Patients with severe internal disease;
* 2. The patients are suffering from gynecologic inflammation or active genital tubercle bacillus;
* 3. The patient has other uterine diseases or the abnormal uterine cavity which can't be restored by surgery;
* 4. Infertility due to a man's cause;
* 5. The patient has a previous history of cancer and is undergoing radiotherapy or chemotherapy;
* 6. HIV positive
* 7. Active hepatitis B or C infection, syphilis seropositive
* 8. Laboratory routine check index abnormality, such as Hb（hemoglobin）<8.0 g/dL,WBC（white blood cell count）<3,000/ml, platelet counts<75 000/mm3, AST（glutamic oxalacetic transaminase）>ULN（upper limit of normal），ALT（Glutamic pyruvic transaminase）>ULN and so on;
* 9. Patients have any complications that may interfere with safety or efficacy or predict life expectancy of less than 24 months;
* 10. Mental illness in the past 6 months;
* 11. Patients have a history of drug or alcohol abuse or dependence in the past two years;
* 12. Unable or unwilling to give informed consent.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
changes of Endometrial thickness | at the 1, 3，6 and 9 months after surgery
  Measure the endometrial thickness during periovulatory period on ultrasound by the same trained medical sonographers at 1,3,6 and 9 months after surgery, comparing with pre-operation.
changes of Menstrual blood volume | at the 1, 3，6 and 9 months after surgery
  Estimate the menstrual blood volume after surgery by the number of sanitary napkins per day and number of days to menstruation at 1, 3, 6, 9 months after surgery, which will be compared with pre-operation.

SECONDARY OUTCOMES:
pregnancy rate | 24 months
  Ultrasound reveals that the fetus had a heart activity

CONTACTS AND LOCATIONS:
Overall Officials: Wang Liang, Principal Investigator — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China